CLINICAL TRIAL: NCT07166796
Title: Tolvaptan Oral Administration Phase I Clinical Trial
Brief Title: a Phase I PK Study in Healthy Male Subjects. 2 Groups of Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Beijing Research Institute (Industry)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-06-801-01
Record Dates: First submitted 2025-08-25; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Health Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single dose (Experimental)
  Interventions: Drug: singe dose 15mg; Drug: single dose 30mg; Drug: single dose 60mg; Drug: single dose 120mg
- multi dose (Experimental)
  Interventions: Drug: multi dose 30mg; Drug: multi dose 60mg

INTERVENTIONS:
Drug: singe dose 15mg — succesfule screened subject, take single dose of 15mg Tolvaptan tablet with no feeding.
  Arms: single dose
Drug: single dose 30mg — succesfule screened subject, take single dose of 30mg Tolvaptan tablet with no feeding.
  Arms: single dose
Drug: single dose 60mg — succesfule screened subject, take single dose of 60mg Tolvaptan tablet with no feeding.
  Arms: single dose
Drug: single dose 120mg — succesfule screened subject, take single dose of 120mg Tolvaptan tablet with no feeding.
  Arms: single dose
Drug: multi dose 30mg — radomize 24 healthy adult male to 2 groups, 12 subjects each. One group take 30mg Tolvaptan. First day, with no feeding, take single 30mg dose, then start from day 3rd, take medication for 7 days. 8 days treatment in total.
  Arms: multi dose
Drug: multi dose 60mg — radomize 24 healthy adult male to 2 groups, 12 subjects each. One group take 60mg Tolvaptan. First day, with no feeding, take single 60mg dose, then start from day 3rd, take medication for 7 days. 8 days treatment in total.
  Arms: multi dose

SUMMARY:
Tolvaptan oral administraction phase I PK clinical trial. Two groups of healthy male subjects. One group receives single dose of Tolvaptan. The other group receives multi dose of Tolvaptan.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers.
2. Aged 18 to 40 years old.
3. Weight no less than 50kg and within the range of standard weight (body mass index between 19 and 24).
4. Auxiliary examinations: blood routine and coagulation, urine routine, blood biochemistry (total protein, albumin, blood glucose, total bilirubin, AST (GOT), ALT (GPT), ALP, γ-GTP, LDH, CK (CPK), total cholesterol, triglycerides, urea nitrogen, creatinine, uric acid, Na, K, Cl, Mg, Ca, P), hepatitis B surface antigen, hepatitis C antibody, HIV antibody, syphilis antibody, 12-lead electrocardiogram, 24-hour ambulatory electrocardiogram (Holter) examination, all items are normal.
5. Signed the informed consent form.

Exclusion Criteria:

1. The patient has a history of heart, liver, kidney, digestive tract, metabolic, respiratory, blood, mental, nervous system and other disorders, and the doctor's judgment is not suitable.
2. Hepatitis B virus, syphilis, hepatitis C virus, HIV infection.
3. Patients with a history of clinically significant arrhythmias of various types, including rapid and slow types, such as atrioventricular block, sinus arrest, and supraventricular tachycardia, were assessed by the investigators.
4. He has a history of postural hypotension (blood pressure drop ≥20/10mmHg when he changes from lying position to standing position, accompanied by dizziness and other symptoms), standing dizziness, collapse, fainting, and vertigo.
5. Quiet for more than 3 minutes, sitting pulse below 55 beats/min or more than 90 beats/min.
6. Quiet for more than 3 minutes, sitting systolic blood pressure is lower than 100mmHg or higher than 140mmHg; Diastolic depression of 60mmHg or higher than 90mmHg.
7. Various voiding disorders (frequent urination, or difficulty urinating, etc.).
8. Have a family history of genetic diseases (including a history of genetically predisposed arrhythmias in relatives).
9. A history, allergy or propensity to be allergic to drugs or any other substance.
10. Smokers, alcoholics, or other drug addicts.
11. Physical examination had clinically significant positive findings.
12. People who have donated blood or been sampled as a subject within the last 3 months.
13. People who have taken prophylactic or therapeutic drugs in the last 2 weeks.
14. Otherwise, the clinical trial physician or the clinical trial physician determines that the safety of the trial is affected.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2006-10-01 (Actual); Primary Completion 2007-01-31 (Actual); Study Completion 2007-01-31 (Actual)

PRIMARY OUTCOMES:
single dose Tolvaptan plasma pharmacokinetics, and its motablics DM-4103 and DM-4107 | Day 1 pre-dose and post-dose 0.5hour, 1 ,2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours
  peak concentration (Cmax)
multi dose Tolvaptan plasma pharmacokinetics and it's motablics DM-4107 and DM-4103 | Day 1 & Day 9 at pre-dose, post-dose 0.5hr, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 (2nd and 10th day) and 48 (day 3rd and 11th). For other dosing day ( day 4 to 8) to collect at pre-dose( 24hr after last dose) point.
  peak concentration (Cmax)
single dose Tolvaptan plasma pharmacokinetics, and its motablics DM-4103 and DM-4107 | Day 1 pre-dose and post-dose 0.5 hour, 1 ,2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours
  time to peak (Tmax)
Tolvaptan plasma pharmacokinetics, and its motablics DM-4103 and DM-4107 | Day 1 pre-dose and post-dose 0.5 hour, 1 ,2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours
  area under the drug-time curve (AUC0-t and AUC0-∞)
single dose Tolvaptan plasma pharmacokinetics, and its motablics DM-4103 and DM-4107 | Day 1 pre-dose and post-dose 0.5 hour, 1 ,2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours
  elimination half-life (t1/2)
single dose Tolvaptan plasma pharmacokinetics, and its motablics DM-4103 and DM-4107 | Day 1 pre-dose and post-dose 0.5 hour, 1 ,2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours
  apparent clearance (CL/F)
single dose Tolvaptan plasma pharmacokinetics, and its motablics DM-4103 and DM-4107 | Day 1 pre-dose and post-dose 0.5 hour, 1 ,2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120 and 144 hours
  apparent volume of distribution (Vd/F)
multi dose Tolvaptan plasma pharmacokinetics and it's motablics DM-4107 and DM-4103 | Day 1 & Day 9 at pre-dose, post-dose 0.5hr, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 (2nd and 10th day) and 48 (day 3rd and 11th). For other dosing day ( day 4 to 8) to collect at pre-dose( 24hr after last dose) point
  time to peak (Tmax)
multi dose Tolvaptan plasma pharmacokinetics and it's motablics DM-4107 and DM-4103 | Day 1 & Day 9 at pre-dose, post-dose 0.5hr, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 (2nd and 10th day) and 48 (day 3rd and 11th). For other dosing day ( day 4 to 8) to collect at pre-dose( 24hr after last dose) point
  area under the drug-time curve (AUC0-t and AUC0-∞)
multi dose Tolvaptan plasma pharmacokinetics and it's motablics DM-4107 and DM-4103 | Day 1 & Day 9 at pre-dose, post-dose 0.5hr, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 (2nd and 10th day) and 48 (day 3rd and 11th). For other dosing day ( day 4 to 8) to collect at pre-dose( 24hr after last dose) point
  elimination half-life (t1/2)
multi dose Tolvaptan plasma pharmacokinetics and it's motablics DM-4107 and DM-4103 | Day 1 & Day 9 at pre-dose, post-dose 0.5hr, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 (2nd and 10th day) and 48 (day 3rd and 11th). For other dosing day ( day 4 to 8) to collect at pre-dose( 24hr after last dose) point
  apparent clearance (CL/F)
multi dose Tolvaptan plasma pharmacokinetics and it's motablics DM-4107 and DM-4103 | Day 1 & Day 9 at pre-dose, post-dose 0.5hr, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36 (2nd and 10th day) and 48 (day 3rd and 11th). For other dosing day ( day 4 to 8) to collect at pre-dose( 24hr after last dose) point
  apparent volume of distribution (Vd/F)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Liu H, Liu T, Liu M, Zheng X, Zhong W, Zhao Q, Jiang J, Hu P, Li Y. Clinical trial on the pharmacokinetics, pharmacodynamics and safety of tolvaptan in healthy Chinese males: an open-label, single and multiple dosage, parallel group study. Front Pharmacol. 2025 Nov 21;16:1713702. doi: 10.3389/fphar.2025.1713702. eCollection 2025. PMID 41357896